CLINICAL TRIAL: NCT05652010
Title: A Randomized, Controlled Clinical Investigation of an Improved Two-piece Stoma Product for People Living With a Stoma
Brief Title: Clinical Investigation of an Improved Two-piece Stoma Product for People Living With a Stoma
Acronym: CP343
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP343
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Surgical Stomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- New coupling (Experimental): The arm includes the new 2-piece coupling
  Interventions: Device: New 2-piece Coupling
- Comparator device (Active Comparator): The arm includes the existing 2-piece coupling
  Interventions: Device: SenSura Mio Click

INTERVENTIONS:
Device: New 2-piece Coupling — Flat or concave baseplate. SenSura Mio Click maxi bag (open, wide outlet) with new 50mm Ø coupling.
  Arms: New coupling
Device: SenSura Mio Click — Flat or concave baseplate. SenSura Mio Click maxi bag (open, wide outlet) with 50mm Ø coupling.
  Arms: Comparator device

SUMMARY:
Open-label, randomized, controlled, comparative, cross-over study with 2 test sequences comparing a new 2-piece coupling system with SenSura Mio Click.

DETAILED DESCRIPTION:
It will be a 1:1 randomization into the two possible treatment sequences

Each test period is 3 weeks (± 2 days), total study period is 6 weeks (± 4 days).

All visits will be performed as remote virtual calls. At the visits, the investigator will give instructions for the coming period and check that the trial is running as planned. At every bag change the subject will be asked to complete a questionnaire.

A follow-up call will be scheduled 7±1 days after each test visit to ensure compliance with the provided product and study procedures. Additional calls may be scheduled if needed.

Minimum 40 participants will be enrolled and randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written consent to participate by signing the Informed Consent Signature Form
2. Be at least 18 years of age and have full legal capacity
3. Is able to handle (apply, remove, cut, etc.) the product and do the assessments themselves
4. Has an ileostomy or colostomy with consistent liquid fecal output (for colostomy: 6-7 Bristol stool scale)
5. Currently use SenSura Mio Click 2p Click flat or concave with 50 mm coupling size
6. Have had their ostomy for at least 90 days
7. Be willing to change the bag at least twice per week
8. Is willing and suitable (determined by the Principal Investigator or designee) to use flat or concave 2p open product during the investigation
9. Is willing to use 2p maxi open bags during the investigation

Exclusion Criteria:

1. Is currently receiving or have within the past 60 days received radio-and/or chemotherapy

   - Low doses radio- and/or chemotherapy (assessed by Principal Investigator) is allowed for indications other than cancer.
2. Is currently receiving or have within the past 30 days received topical steroid treatment in the peristomal skin area, e.g., lotion or spray

   * Low dose systemic steroid treatment (e.g., inhalation) assessed by the investigator are allowed.
   * Other systemic steroid treatment (e.g., injection or tablet) are not allowed.
3. Is pregnant and/or breast-feeding
4. Have a loop ileostomy
5. Is currently using convex baseplate
6. Has known hypersensitivity towards any of the products used in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selwyn Spangenthal, MD, Principal Investigator — American Health Research
Locations (1):
- American Health Research, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 15 Feb 2023 Last Patient Out: 17 July 2023
Pre-assignment Details: 51 participants were enrolled. After enrolment, one participant was excluded due to meeting exclusion crit. 5. Three participants wished to discontinue before randomization. Therefore, only 47 started in the treatment arms, while the safety population was 51.
Groups:
- New Coupling First, Then Comparator Device: Cross-over study: First intervention (3 weeks), followed by Second intervention (3 weeks).
- Comparator Device First, Then New Coupling: Cross-over study: First intervention (3 weeks), followed Second intervention (3 weeks).
Period: First Intervention
Arm/Group | New Coupling First, Then Comparator Device | Comparator Device First, Then New Coupling
Started | 22 | 25
Completed | 22 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | New Coupling First, Then Comparator Device | Comparator Device First, Then New Coupling
Started | 22 | 24
Completed | 21 | 24
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographics are described for the total ITT population
Groups:
- All Participants: Demographics are described for the total Intention-to-Treat (ITT) population
Arm/Group | All Participants
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Stoma type [Count of Participants; unit: Participants]
  Colostomy | 19
  Ileostomy | 28

OUTCOME MEASURES:

1. Primary Outcome: Leakage Through Coupling Registered at Each Bag Change (Yes/no)
Description: Output visible inside and/or outside the coupling system when the bag is changed.
  Presented in proportion of bag changes (with leakage) per participant.
Time Frame: 3 weeks
Population: ITT
Measure: Mean (95% Confidence Interval); unit: Proportion of bag changes/participant
Groups:
- New Coupling: Both test sequences with new coupling
- Comparator Device: Both test sequences with comparator device
Arm/Group | New Coupling | Comparator Device
Number analyzed (Participants) | 45 | 46
Proportion of bag changes/participant | 0.151 [0.089 to 0.247] | 0.237 [0.156 to 0.341]
Statistical Analysis 1: Comparison: New Coupling vs Comparator Device; Test type: Other — Comparative study; p = 0.164, Mixed Models Analysis — P=0.164 for testing the hypothesis that OR=1; Generalized linear mixed model. As it was an exploratory study no adjustment for multiple comparison was performed; Odds Ratio (OR) = 0.576, 95% CI 2-sided [0.2634 to 1.2659] — P=0.164 for testing the hypothesis that OR=1

2. Secondary Outcome: How Satisfied Are You With the New Coupling?
Description: Satisfaction with new coupling evaluated at end of study by a question on a 4-point scale (very satisfied - satisfied - dissatisfied - very dissatisfied)
Time Frame: 3 weeks - evaluated at the end of the study
Measure: Count of Participants; unit: Participants
Groups:
- Very Satisfied / Satisfied: The number of participants that selected very satisfied or satisfied
- Dissatisfied / Very Dissatisfied: The number of participants that selected very dissatisfied or very dissatisfied
Arm/Group | Very Satisfied / Satisfied | Dissatisfied / Very Dissatisfied
Number analyzed (Participants) | 39 | 39
Participants | 35 | 4
Statistical Analysis 1: Comparison: Very Satisfied / Satisfied vs Dissatisfied / Very Dissatisfied; Test type: Other; p < 0.0001, Exact test in the binomial distribution; Exact test in the binomial distribution tested if the proportion of very satisfied/satisfied was sign. different from 50% when using a 5% test level; Binominal = 0.90, 95% CI 2-sided [0.75 to 0.97] — The binomial proportion is based on subjects that have answered the questions. Exact test in the binomial distribution

3. Secondary Outcome: Would You Consider Using the New Coupling in the Future?
Description: Preference evaluated at end of the investigation by the question "Would you consider using the new coupling in the future?" (Yes/No)
Time Frame: Based on 3 weeks - evaluated at the end of the study period
Measure: Count of Participants; unit: Participants
Groups:
- Would Consider Using the New Coupling in the Future: Yes: The number of participants that would consider using the new coupling in the future
- Would Consider Using the New Coupling in the Future: No: The number of participants who would not consider using the new coupling in the future
Arm/Group | Would Consider Using the New Coupling in the Future: Yes | Would Consider Using the New Coupling in the Future: No
Number analyzed (Participants) | 39 | 39
Participants | 32 | 7
Statistical Analysis 1: Comparison: Would Consider Using the New Coupling in the Future: Yes vs Would Consider Using the New Coupling in the Future: No; Test type: Other — The binomial proportion is based on subjects that have answered the questions. Exact test in the binomial distribution; p < 0.0001, Exact test in the binominal distribution; Exact test in the binomial distribution tested if the proportion of YES was significantly different from 50% when using a 5% test level; Binominal = 0.82, 95% CI 2-sided [0.66 to 0.92]

4. Post Hoc Outcome: Leakage Visible Outside the Coupling
Description: Leakage from coupling, visible outside coupling on baseplate when the bag is changed.
  Presented in proportion of bag changes (with leakage) per participant.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: Proportion of bag changes/participant
Arm/Group | New Coupling | Comparator Device
Number analyzed (Participants) | 45 | 46
Proportion of bag changes/participant | 0.012 [0.004 to 0.032] | 0.044 [0.024 to 0.082]
Statistical Analysis 1: Comparison: New Coupling vs Comparator Device; Test type: Other; p = 0.027, Mixed Models Analysis — P=0.027 for testing the hypothesis that OR=1; Generalized linear mixed model; Odds Ratio (OR) = 0.259, 95% CI 2-sided [0.078 to 0.855] — P=0.027 for testing the hypothesis that OR=1

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the study period of 6 weeks.
Arm/Group | New Coupling | Comparator Device
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 1/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Coupling (N=47) | Comparator Device (N=47)
Skin breakdown around peristomal area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Baseplate used prior to randomization was deep convex (exclusion criterium #5). This led to leakage due to improper fit. Subject was withdrawn.

LIMITATIONS AND CAVEATS:
The investigation was non-blinded. However, the two products came from the same manufacturer and were very similar in appearance.

Subjects were instructed to register leakage through the coupling seen from the outside before opening the coupling. However, the accompanying instructive drawings showed leakage in an opened coupling, which could have resulted in overreporting of leakages that would only be visible after opening or happening when opening the coupling.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT05652010/Prot_SAP_000.pdf